CLINICAL TRIAL: NCT04327089
Title: An Open-Label Phase 1 Study to Evaluate the Pharmacokinetics and Drug-Drug Interactions of Setanaxib in Healthy Adult Male and Female Subjects
Brief Title: Study to Evaluate the Pharmacokinetics and Drug-Drug Interactions of Setanaxib in Healthy Adult Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calliditas Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GSN000310
Record Dates: First submitted 2020-03-12; First posted 2020-03-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2021-05

CONDITIONS: Phase 1
MeSH Terms: interventions — setanaxib

STUDY DESIGN:
Intervention Model Description: Open-Label Phase 1 Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1- Cohort 1 (Experimental): Single oral dose of 400 mg Setanaxib administered as 1x400 mg tablet in fasting conditions.
  Interventions: Drug: Setanaxib
- Part 1- Cohort 2 (Experimental): Single oral dose of 800 mg Setanaxib administered as 2x400 mg tablet in fasting conditions.
  Interventions: Drug: Setanaxib
- Part 1- Cohort 3 (Experimental): Single oral dose of 1200 mg Setanaxib administered as 3x400 mg tablet in fasting conditions.
  Interventions: Drug: Setanaxib
- Part 1- Cohort 4 (Experimental): Single oral dose of 1600 mg Setanaxib administered as 4x400 mg tablet in fasting conditions.
  Interventions: Drug: Setanaxib
- Part 2- Cohort 5 (Experimental): Repeated 10-Day dosing of 1200mg/day of Setanaxib administered as 2x400mg tablet in the morning and as 1x400mg tablet in the evening in fedding conditions.
  Interventions: Drug: Setanaxib
- Part 2- Cohort 6 (Experimental): Repeated 10-Day dosing of 1600mg/day of Setanaxib administered as 2x400mg tablet in the morning and as 2x400mg tablet in the evening in fedding conditions.
  Interventions: Drug: Setanaxib
- Cohort 7 (Experimental): Repeated 10-Day dosing of 1600mg/day of Setanaxib administered as 2x400mg tablet in the morning and as 2x400mg tablet in the evening in fedding conditions. Additionnaly, this cohort includes the evaluation of potential Drug-Drug interactions with CYPs and transporters.
  Interventions: Drug: Setanaxib

INTERVENTIONS:
Drug: Setanaxib — Nox 1/4 inhibitor
  Other Names: GKT137831

SUMMARY:
The study is a monocentric, open label, phase 1 study to evaluate the pharmacokinetics, and in particular the dose proportionality of setanaxib and its metabolites after a single oral dose (400 mg, 800 mg, 1200 mg, and 1600 mg) (Part 1) and after multiple oral doses (Part 2).

DETAILED DESCRIPTION:
The study is a monocentric, open label, phase 1 study to evaluate the pharmacokinetics, and in particular the dose proportionality of setanaxib and its metabolites after a single oral dose (400 mg, 800 mg, 1200 mg, and 1600 mg) (Part 1) and after multiple oral doses (Part 2). The study will include 2 parts conducted in separate cohorts of subjects.

* Part 1 of the study will be an open label, single dose study evaluating the pharmacokinetics, and in particular the dose proportionality of setanaxib formulated as tablets, in 4 separate cohorts of 6 to 8 healthy adult subjects
* Part 2 of the study will assess the pharmacokinetics of setanaxib tablets, expand the evaluation of potential drug-drug interactions, and assess the safety of setanaxib tablets at doses up to 1600mg/day for 14 days in separate 2 cohorts. The evaluation of drug-drug interactions will be carried out only at the top dose. Accordingly, a larger cohort (i.e. 16 subjects) will be included in Cohort 7.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female aged 18 to 49 years
2. Provision of written informed consent to participate as shown by a signature on the subject consent form
3. Smoke no more than 5 cigarettes a day are permitted. Smocking (including the use of smocking substitute e.g. nicotine patch) is not permitted from screening to the end of study visit
4. Body weight of at least 45kg and a BMI included between 18.0 and 35.0 kg/m2
5. Female subjects of childbearing potential must use a highly effective method of contraception to prevent pregnancy for 4 weeks before inclusion and must agree to continue strict contraception for 30 days after last administration of IMP. Male participants with female partners of childbearing potential must be willing to use a condom and require their partner to use an additional form of adequate contraception as approved by the Investigator. This requirement begins at the time of informed consent and ends at least 3 months after the last administration of IMP. Male study participants must also not donate sperm from baseline until 3 months after the last administration of IMP.
6. Considered as healthy after a comprehensive clinical assessment (detailed medical history and complete physical examination)
7. Normal Blood Pressure (BP) and Heart Rate (HR) at the screening visit after 10 minutes in supine position.
8. Normal ECG recording on a 12-lead ECG at the screening visit:
9. Laboratory parameters within the normal range of the laboratory (hematological, blood chemistry tests, urinalysis). Individual values out of the normal range can be accepted if judged non-clinically significant by the Investigator
10. Has not consumed and agrees to abstain from taking any dietary supplements or non-prescription drugs over the 7 days prior to screening.
11. Has not consumed and agrees to abstain from taking any prescription drugs except contraception.
12. Has not consumed alcohol containing beverages over the 48 hours prior to hospitalization
13. Has not consumed grapefruit or grapefruit juice over the 48 hours prior to hospitalization
14. Has the ability to understand the requirements of the study and is willing to comply with all study procedures
15. Registered with the French Social Security in agreement with the French law on biomedical experimentation and register to the "Fichier national des personnes qui se prêtent à des recherches biomédicales"

Exclusion Criteria:

1. Have already received setanaxib
2. Contraindication(s) for any of the substrates used in the study
3. Any history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic or infectious disease
4. Any history of severe cardiovascular disease, and any personal or family history of long QT syndrome, or evidence of abnormalities in cardiac conduction
5. Frequent headaches and / or migraine, recurrent nausea and / or vomiting
6. Symptomatic hypotension whatever the decrease of blood pressure or asymptomatic postural hypotension defined by a decrease in SBP or DBP equal to or greater than 20 mmHg within two minutes when changing from the supine to the standing position
7. Blood donation (including in the frame of a clinical study) within 2 months before administration;
8. General anesthesia within 3 months before administration
9. Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician
10. Inability to abstain from intensive muscular effort
11. No possibility of contact in case of emergency
12. Any drug intake (except paracetamol or oral contraception) during the last month prior to the first administration
13. History or presence of drug or alcohol abuse (alcohol consumption > 40 grams / day)
14. Excessive consumption of beverages with xanthine bases (> 4 cups or glasses / day) during the last 30 days
15. Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests
16. Positive results of screening for drugs of abuse
17. Any contraindication to the administration of midazolam, adefovir, losartan, omeprazole, sitagliptin
18. Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development
19. Currently in exclusion period from a previous study
20. Administrative or legal supervision
21. Subject who would receive more than 4500 euros as indemnities for his participation in biomedical study within the 12 last months, including the indemnities for the present study.
22. Minor, pregnant or breast-feeding women, persons deprived of liberty by judicial or administrative decision, persons receiving psychiatric care and persons admitted to a health or social institution, adult subject to legal protection or unable to express consent.
23. Positive results for SARS-CoV-2 tests.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Dose proportionality of setanaxib tablets after single oral administration of different doses. | 144 hours
  Measure the AUC and bioavailability (particularly the dose proportionality) of setanaxib tablets, after single oral administration of different doses (400, 800, 1200 and 1600mg) in healthy adult male and female subjects.
Drug-drug interactions of multiple oral administrations of setanaxib with 5 drugs that interact with CYP3A4, OAT1, OAT3, 2C9 and 2C19. | 14 days
  Measure the changes in AUC of 5 drugs that interact with CYP3A4, OAT1, OAT3, 2C9 and 2C19 in healthy adult male (8) and female (8) subjects after multiple administrations of Setanaxib at dose of 1600mg only (cohort 6) or 800mg (cohort 7).
Assessment of safety after multiple oral administration of different doses of setanaxib. | 10 days
  To evaluate the biological, physiological and treatment-related adverse events of setanaxib after multiple oral administration doses up to 1600 mg/day in healthy male and female subjects.

SECONDARY OUTCOMES:
Assessment of safety after single oral administration of different doses of setanaxib. | 144 hours
  To evaluate the biological, physiological and treatment-related adverse events of setanaxib tablets after single oral administration of 4 different doses in healthy male and female subjects.
Dose proportionality of setanaxib tablets after multiple oral administration of different doses. | 10 days
  Measure the AUC and bioavailability (particularly the dose proportionality) of setanaxib tablets after multiple oral administration at 2 different doses in healthy adult male and female subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Optimed, Gières, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gage MC, Thippeswamy T. Inhibitors of Src Family Kinases, Inducible Nitric Oxide Synthase, and NADPH Oxidase as Potential CNS Drug Targets for Neurological Diseases. CNS Drugs. 2021 Jan;35(1):1-20. doi: 10.1007/s40263-020-00787-5. Epub 2021 Jan 30. PMID 33515429